CLINICAL TRIAL: NCT02038777
Title: A PHASE 1 STUDY TO EVALUATE THE SAFETY, TOLERABILITY, EFFICACY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF PF-04449913 (GLASDEGIB), AN ORAL HEDGEHOG INHIBITOR, ADMINISTERED AS A SINGLE AGENT IN JAPANESE PATIENTS WITH SELECT HEMATOLOGIC MALIGNANCIES AND IN COMBINATION WITH INTENSIVE CHEMOTHERAPY, LOW-DOSE ARA-C, OR AZACITIDINE IN PATIENTS WITH ACUTE MYELOID LEUKEMIA OR HIGH-RISK MYELODYSPLASTIC SYNDROME
Brief Title: A Study Of PF-04449913 In Japanese Patients With Select Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B1371005; NCT02038777 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2014-01-14; First posted 2014-01-17 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Hematologic Malignancies
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Neoplasms | interventions — glasdegib; Cytarabine; Daunorubicin; Azacitidine

STUDY DESIGN:
Intervention Model Description: MTD was determined in monotherapy cohort. Then two combination cohorts (Combination Cohorts 1 and 2) were added to evaluate the safety of glasdegib administered with chemotherapies. Another combination cohort (Combination Cohort 3) was added to evaluate the safety of glasdegib administered with Azacitidine. Then, Continuation Cohort which allows one Japanese patient enrolled from another trial in the same project was added. Afther that, Expansion Cohort of LDAC Combination for efficacy was added.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Monotherapy Cohort (Experimental): PF-04449913 Monotherapy
  Interventions: Drug: PF-04449913
- Combination Cohort 1 (Experimental): PF-04449913 in combination with low dose ARA-C (LDAC)
  Interventions: Drug: PF-04449913; Drug: Low dose ARA-C (LDAC)
- Combination Cohort 2 (Experimental): PF-04449913 in combination with intensive chemotherapy: PF-04449913 administered continuously for 28 days. Daunorubicin given using 60 mg/m2 for 3-days together with cytarabine 100 mg/m2 on days 1 through 7 followed by cytarabine 1g/m2 on days 1, 3, and 5 during 2-4 cycles of consolidation therapy.
  Interventions: Drug: PF-04449913; Drug: Daunorubicin; Drug: Cytarabine
- Azacitidine Combination Cohort (Experimental): PF-04449913 in combination with azacitidine
  Interventions: Drug: PF-04449913; Drug: Azacitidine
- Continuation Cohort (Experimental): PF-04449913 Monotherapy for one patient rolled-over from another trial in the same project.
  Interventions: Drug: PF-04449913
- Expansion Cohort of LDAC Combination for Efficacy (Experimental): PF-04449913 in combination with LDAC to evaluate efficacy
  Interventions: Drug: PF-04449913; Drug: LDAC

INTERVENTIONS:
Drug: PF-04449913 — PF-04449913 administered orally and continuously in 28 day cycles.
  Arms: Continuation Cohort; Monotherapy Cohort
Drug: PF-04449913 — PF-04449913 administered orally and continuously in 28 day cycles.
  Arms: Combination Cohort 1
Drug: Low dose ARA-C (LDAC) — Low dose ARA-C (LDAC) administered at 20 mg SQ, BID on Days 1 through 10.
  Arms: Combination Cohort 1
Drug: PF-04449913 — PF-04449913 administered orally and continuously in 28 day cycles.
  Arms: Combination Cohort 2
Drug: Daunorubicin — Daunorubicin given using 60 mg/m2 for 3-days.
  Arms: Combination Cohort 2
Drug: Cytarabine — Cytarabine 100 mg/m2 on days 1 through 7.
  Arms: Combination Cohort 2
Drug: PF-04449913 — PF-04449913 administered orally and continuously in 28 day cycles.
  Arms: Azacitidine Combination Cohort
Drug: Azacitidine — Azacitidine Combination Cohort; Azacitidine 75 mg/m2 for 7 days.
  Arms: Azacitidine Combination Cohort
Drug: PF-04449913 — PF-04449913 administered orally and continuously in 28 day cycles.
  Arms: Expansion Cohort of LDAC Combination for Efficacy
Drug: LDAC — Low dose ARA-C (LDAC) administered at 20 mg SQ, BID on Days 1 through 10.
  Arms: Expansion Cohort of LDAC Combination for Efficacy

SUMMARY:
This is an open-label, multi-center, Phase 1 study of PF-04449913 in Japanese patients. PF-04449913 will be administered orally as a single agent in patients with select advanced hematologic malignancies, or in combination with LDAC [Low-Dose Ara-C] or cytarabine and daunorubicin in previously untreated patients with AML [Acute Myeloid Leukemia] or high-risk MDS [Myelodysplastic Syndrome], or in combination with azacitidine in previously untreated patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients with select advanced hematologic malignancies who are refractory, resistant or intolerant to prior therapies for monotherapy cohort.
* Patients with AML or High-Risk MDS who are newly diagnosed and previously untreated for combination cohort.
* Patients with AML who are newly diagnosed and previously untreated for azacitidine combination cohort.
* ECOG [Eastern Cooperative Oncology Group] performance status 0 to 2
* Adequate organ function

Exclusion Criteria:

* Patients with active CNS disease
* Patient with active malignancy with the exception of basal cell carcinoma, non melanoma skin cancer, carcinoma in situ cervical
* Patient has an active, life threatening or clinically significant uncontrolled systemic infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Japan (9):
  - Japanese Red Cross Nagoya First Hospital, Nagoya, Aichi-ken
  - Kobe University Hospital, Kobe, Hyōgo
  - Tohoku University Hospital, Sendai, Miyagi
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Akita University Hospital, Akita
  - Kyushu University Hospital, Fukuoka
  - Tokyo Medical University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371005&StudyName=A%20Study%20Of%20PF-04449913%20In%20Japanese%20Patients%20With%20Select%20Hematologic%20Malignancies

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 54 participants signed the inform consent form (ICF). Out of which 6 participants were screen failure, 48 actually enrolled into the study and assigned to study treatment. One participant was randomized but not treated.
Groups:
- Monotherapy Cohort: PF-04449913 (Glasdegib) 25 mg: Participants with advanced hematologic malignancies received PF-04449913 25 milligram (mg) tablets orally, a single dose on Day -5 of Cycle 1 and then continuously once daily (QD) from Cycle 1/Day 1 in 28-day cycles, maximum up to 12 cycles or until disease progression or relapse, or participant withdrawal, or unacceptable toxicity (whichever occurred first).
- Monotherapy Cohort: PF-04449913 50 mg: Participants with advanced hematologic malignancies received PF-04449913 50 mg tablets orally, a single dose on Day -5 of Cycle 1 and then continuously QD from Cycle 1/Day 1 in 28-day cycles, maximum up to 12 cycles or until disease progression or relapse, or participant withdrawal, or unacceptable toxicity (whichever occurred first).
- Monotherapy Cohort: PF-04449913 100 mg: Participants with advanced hematologic malignancies received PF-04449913 100 mg tablets orally, a single dose on Day -5 of Cycle 1 and then continuously QD from Cycle 1/Day 1 in 28-day cycles, maximum up to 12 cycles or until disease progression or relapse, or participant withdrawal, or unacceptable toxicity (whichever occurred first).
- Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg: Participants with previously untreated acute myeloid leukemia (AML)/high-risk myelodysplastic syndrome (MDS) and unfit for intensive chemotherapy, received PF-04449913 100 mg tablets continuously QD from Cycle 1/Day 3 in 28 day cycles and low dose Ara-cytarabine (LDAC) 20 mg was administered subcutaneously (SC) twice daily for first 10 days of the 28-day cycles, maximum up to up to 12 cycles or until disease progression or relapse, or participant refusal, or unacceptable toxicity occurs (whichever occurred first).
- Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin: Participants with previously untreated AML/high-risk MDS and fit for intensive chemotherapy, participants started receiving PF-04449913 100 mg tablets QD from Day -3 up to Day 28 for first induction cycle and then continuously QD from Cycle 1/Day 1 in 28 day cycles for rest of treatment duration along with Cytarabine 100 mg per square meter (mg/m^2) was administered daily by continuous intravenous (IV) infusion for first 7 days of Cycle and Daunorubicin 60 mg/m^2 daily IV for first 3 days of Cycle. Participants with <= 5% bone marrow blasts had second cycle of induction. Participants achieving a complete response after the completion of induction therapy were eligible to begin consolidation cycles. During consolidation, participants received PF-04449913 100 mg tablets orally QD in 28 day cycle along with Cytarabine 1g/m^2 QD on Day 1, 3 and 5 of 28 day cycle. Consolidation was of 2 to 4 cycles. Post-consolidation participants received PF-04449913 100 mg tablets orally QD in 28-day cycle for maintenance up to maximum of 6 cycles.
- Combination Cohort 3: PF-04449913 100 mg + Azacitidine: Participants with untreated AML and eligible for non-intensive chemotherapy received PF-04449913 100 mg tablets orally, continuously QD from Cycle 1/Day 2 in 28 day cycles along with azacitidine 75 mg/m^2/day SC or IV daily on Days 1-7 of each 28-day cycle. Treatment continued for at least 6 cycles, or until disease progression or relapse, or participant withdrawal, or unacceptable toxicity, or death (whichever occurred first).
- Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg: Participants with myelofibrosis treated with PF-04449913 in B1371013 received the same dose (100 mg) of PF-04449913 as at the time of discontinuation from study B1371013 from Cycle 1/Day 1 until disease progression or relapse, or participant withdrawal, or unacceptable toxicity, or death (whichever occurred first).
- Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg: Participants with previously untreated AML or high-risk MDS and unfit for intensive chemotherapy received PF-04449913 100 mg tablets continuously QD from Cycle 1/Day 1 in 28-day cycles and LDAC 20 mg SC twice daily for first 10 days of the 28-day cycles, until disease progression or relapse, or participant withdrawal, or unacceptable toxicity, or death (whichever occurred first).
Period: Overall Study
Arm/Group | Monotherapy Cohort: PF-04449913 (Glasdegib) 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin | Combination Cohort 3: PF-04449913 100 mg + Azacitidine | Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Started | 3 | 5 | 6 | 6 | 6 | 6 | 1 | 15
Treated (Safety Set) | 3 | 4 | 6 | 6 | 6 | 6 | 1 | 15
Completed | 2 | 1 | 3 | 2 | 3 | 2 | 0 | 3
Not Completed | 1 | 4 | 3 | 4 | 3 | 4 | 1 | 12
Not completed — Death | 0 | 2 | 0 | 1 | 2 | 4 | 0 | 11
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Started Chemotherapy | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — participation terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Groups:
- Monotherapy Cohort: PF-04449913 (Glasdegib) 25 mg: Participants with advanced hematologic malignancies received PF-04449913 25 mg tablets orally, a single dose on Day -5 of Cycle 1 and then continuously QD from Cycle 1/Day 1 in 28-day cycles, maximum up to 12 cycles or until disease progression or relapse, or participant withdrawal, or unacceptable toxicity (whichever occurred first).
- Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg: Participants with previously untreated AML/high-risk MDS and unfit for intensive chemotherapy, received PF-04449913 100 mg tablets continuously QD from Cycle 1/Day 3 in 28- day cycles and LDAC 20 mg was administered SC BID for first 10 days of the 28-day cycles, maximum up to up to 12 cycles or until disease progression or relapse, or participant refusal, or unacceptable toxicity occurs (whichever occurred first).
- Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin: Participants with previously untreated AML/high-risk MDS and fit for intensive chemotherapy, participants started receiving PF-04449913 100 mg tablets QD from Day -3 up to Day 28 for first induction cycle and then continuously QD from Cycle 1/Day 1 in 28 day cycles for rest of treatment duration along with Cytarabine 100 mg/m^2 was administered daily by continuous IV infusion for first 7 days of Cycle and Daunorubicin 60 mg/m^2 daily IV for first 3 days of Cycle. Participants with <= 5% bone marrow blasts had second cycle of induction. Participants achieving a complete response after the completion of induction therapy were eligible to begin consolidation cycles. During consolidation, participants received PF-04449913 100 mg tablets orally QD in 28-day cycle along with Cytarabine 1g/m^2 QD on Day 1, 3 and 5 of 28 day cycle. Consolidation was of 2 to 4 cycles. Post-consolidation participants received PF-04449913 100 mg tablets orally QD in 28-day cycle for maintenance up to maximum of 6 cycles.
- Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg: Participants with previously untreated AML or high-risk MDS and unfit for intensive chemotherapy received PF-04449913 100 mg tablets continuously QD from Cycle 1/Day 1 in 28-day cycles and LDAC 20 mg SC twice daily for first 10 days of the 28 day cycles, until disease progression or relapse, or participant withdrawal, or unacceptable toxicity, or death (whichever occurred first).
- Total: Total of all reporting groups
Arm/Group | Monotherapy Cohort: PF-04449913 (Glasdegib) 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin | Combination Cohort 3: PF-04449913 100 mg + Azacitidine | Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg | Total
Number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 6 | 1 | 15 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (9.07) | 67.3 (3.59) | 70 (8.53) | 71.8 (8.73) | 68 (4.94) | 74.5 (6.92) | 77.0 (NA) — Standard deviation could not be estimated as there was only 1 participant evaluable. | 77.5 (5.21) | 72.2 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 1 | 2 | 2 | 1 | 7 | 18
  Male | 2 | 3 | 3 | 5 | 4 | 4 | 0 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 6 | 6 | 6 | 6 | 1 | 15 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 6 | 6 | 6 | 6 | 1 | 15 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs): Monotherapy Cohort
Description: Criteria: Grade >=3 non-hematologic toxicity (nht), except Grade >=3 infection, fever (including febrile neutropenia), infusion related AEs, electrolyte abnormalities, alanine aminotransferase (AT)/aspartate AT elevation that returned to Grade <=1/baseline within 7 days, allergic reactions possibly related to PF-04449913 that led to discontinuation of study drug; Prolonged myelosuppression lasted >42 days from point of detection = absolute neutrophil count < 500/microliter or platelet count <10*10^9/L with a normal bone marrow (<5% blasts and no evidence of disease or dysplasia); Inability to deliver >=80% of the planned study doses for all agents in a combination due to nht; Delay of >28 days in receiving next scheduled cycle due to persisting nht; Asymptomatic participant with Grade >=3 QTc prolongation required repeat testing, re-evaluation by qualified person, and correction of reversible causes for confirmation. Post-correction, if Grade 3 prolongation persisted, event was a DLT.
Time Frame: Day -5 up to Day 28 of Cycle 1 (33 days)
Population: DLT evaluable analysis set included all enrolled participants who received at least 1 dose of study medication and who did not have major treatment deviations during first cycle (DLT observation period).
Measure: Count of Participants; unit: Participants
Groups:
- Monotherapy Cohort: PF-04449913 25 mg: Participants with advanced hematologic malignancies received PF-04449913 25 mg tablets orally, a single dose on Day -5 of Cycle 1 and then continuously QD from Cycle 1/Day 1 in 28-day cycles, maximum up to 12 cycles or until disease progression or relapse, or participant withdrawal, or unacceptable toxicity (whichever occurred first).
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, Treatment Related TEAEs, Grade 3 or 4 TEAEs Based on NCI CTCAE v4.0: Monotherapy Cohort
Description: AE:any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Serious AE:any untoward medical occurrence at any dose that resulted in death;was life threatening;required inpatient hospitalization or prolongation of existing hospitalization;resulted in persistent or significant disability/incapacity;resulted in congenital anomaly/birth defect. TEAEs:events absent before treatment or that worsened relative to pretreatment state. Treatment-related TEAE:any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to drug was assessed by the Investigator. National cancer institute common terminology criteria (NCI-CTCAE) Grade(G) v4.0:G 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; G 4:life-threatening consequence, urgent intervention indicated.
Time Frame: Day 1 up to 28 days after last dose of study drug (For 25 mg: maximum up to 136 days; For 50 mg: maximum up to 179 days; For 100 mg: maximum up to 472 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Participants
  TEAEs | 3 | 4 | 6
  Serious TEAEs | 1 | 3 | 1
  Treatment related TEAEs | 1 | 3 | 5
  Grade 3 or 4 TEAEs | 2 | 1 | 3

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs Abnormalities: Monotherapy Cohort
Description: Vital signs included blood pressure (sitting or supine) and heart rate. Clinically significant changes in vital signs were determined by the investigator's discretion.
Time Frame: For 25 mg: Baseline up to maximum 108 days; For 50 mg: Baseline up to maximum 151 days; For 100 mg: Baseline up to maximum 444 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Worst On-study Laboratory Abnormalities: Monotherapy Cohort
Description: Laboratory parameters included- hematology: lymphocytes/leukocytes percentage (%), neutrophils/leukocytes, basophils/leukocytes, eosinophils/leukocytes and monocytes/leukocytes (%), prothrombin time second (sec), blasts/leukocytes (%); clinical chemistry: lactate dehydrogenase units per liter (u/l), protein gram/liter (g/l), blood urea nitrogen (BUN) millimoles per liter (mmol/l), urate, chloride, calcium (mmol/l); urinalysis: specific gravity, pH, urine glucose and ketones (scalar), nitrite, leukocyte esterase, urine erythrocytes (scalar), urine leukocytes (scalar). In this outcome measure participants for each laboratory parameter were evaluated as normal, abnormal low, abnormal high or abnormal low and an abnormal high. Laboratory values were as per laboratory normal ranges. Values above normal range = abnormal high and below range = abnormal low. Participants with both an abnormal low and high value while on study were reported as 'Abnormal low and Abnormal high'.
Time Frame: For 25 mg: Baseline up to maximum 136 days; For 50 mg: Baseline up to maximum 179 days; For 100 mg: Baseline up to maximum 472 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication. Here, "number of participants analyzed" signifies participants evaluable for the specific parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Participants
  Lymphocytes/Leukocytes: Normal | 0 | 0 | 0
  Lymphocytes/Leukocytes: Abnormal low only | 2 | 4 | 2
  Lymphocytes/Leukocytes: Abnormal high only | 1 | 0 | 2
  Lymphocytes/Leukocytes: Abnormal low and abnormal high | 0 | 0 | 2
  Neutrophils/Leukocytes: Normal | 0 | 0 | 0
  Neutrophils/Leukocytes: Abnormal low only | 2 | 3 | 4
  Neutrophils/Leukocytes: Abnormal high only | 1 | 1 | 1
  Neutrophils/Leukocytes: Abnormal low and abnormal high | 0 | 0 | 1
  Basophils/Leukocytes: Normal | 3 | 2 | 2
  Basophils/Leukocytes: Abnormal low only | 0 | 0 | 0
  Basophils/Leukocytes: Abnormal high only | 0 | 2 | 4
  Basophils/Leukocytes: Abnormal low and abnormal high | 0 | 0 | 0
  Eosinophils/Leukocytes: Normal | 3 | 2 | 4
  Eosinophils/Leukocytes: Abnormal low only | 0 | 1 | 0
  Eosinophils/Leukocytes: Abnormal high only | 0 | 0 | 2
  Eosinophils/Leukocytes: Abnormal low and abnormal high | 0 | 1 | 0
  Monocytes/Leukocytes: Normal | 2 | 0 | 0
  Monocytes/Leukocytes: Abnormal low only | 1 | 2 | 3
  Monocytes/Leukocytes: Abnormal high only | 0 | 2 | 3
  Monocytes/Leukocytes: Abnormal low and abnormal high | 0 | 0 | 0
  Prothrombin time: number analyzed (Participants) | 1 | 4 | 6
  Prothrombin time: Normal | 0 | 0 | 3
  Prothrombin time: Abnormal low only | 0 | 0 | 0
  Prothrombin time: Abnormal high only | 1 | 4 | 3
  Prothrombin time: Abnormal low and abnormal high | 0 | 0 | 0
  Blasts/Leukocytes: number analyzed (Participants) | 0 | 0 | 3
  Blasts/Leukocytes: Normal | 0 | 0 | 1
  Blasts/Leukocytes: Abnormal low only | 0 | 0 | 0
  Blasts/Leukocytes: Abnormal high only | 0 | 0 | 2
  Blasts/Leukocytes: Abnormal low and abnormal high | 0 | 0 | 0
  Lactate dehydrogenase: Normal | 0 | 0 | 1
  Lactate dehydrogenase: Abnormal low only | 0 | 0 | 0
  Lactate dehydrogenase: Abnormal high only | 3 | 4 | 5
  Lactate dehydrogenase: Abnormal low and abnormal high | 0 | 0 | 0
  Protein: Normal | 1 | 0 | 2
  Protein: Abnormal low only | 2 | 3 | 3
  Protein: Abnormal high only | 0 | 1 | 1
  Protein: Abnormal low and abnormal high | 0 | 0 | 0
  BUN: Normal | 0 | 3 | 4
  BUN: Abnormal low only | 1 | 0 | 0
  BUN: Abnormal high only | 2 | 1 | 2
  BUN: Abnormal low and abnormal high | 0 | 0 | 0
  Urate: Normal | 0 | 1 | 2
  Urate: Abnormal low only | 2 | 0 | 0
  Urate: Abnormal high only | 0 | 3 | 4
  Urate: Abnormal low and abnormal high | 1 | 0 | 0
  Chloride: Normal | 2 | 3 | 3
  Chloride: Abnormal low only | 0 | 1 | 1
  Chloride: Abnormal high only | 1 | 0 | 2
  Chloride: Abnormal low and abnormal high | 0 | 0 | 0
  Calcium: Normal | 0 | 2 | 2
  Calcium: Abnormal low only | 3 | 2 | 4
  Calcium: Abnormal high only | 0 | 0 | 0
  Calcium: Abnormal low and abnormal high | 0 | 0 | 0
  Urine specific gravity: Normal | 2 | 3 | 3
  Urine specific gravity: Abnormal low only | 0 | 1 | 3
  Urine specific gravity: Abnormal high only | 1 | 0 | 0
  Urine specific gravity: Abnormal low and abnormal high | 0 | 0 | 0
  Urine pH: Normal | 2 | 3 | 4
  Urine pH: Abnormal low only | 0 | 0 | 0
  Urine pH: Abnormal high only | 1 | 1 | 2
  Urine pH: Abnormal low and abnormal high | 0 | 0 | 0
  Urine glucose: number analyzed (Participants) | 2 | 2 | 4
  Urine glucose: Normal | 2 | 2 | 4
  Urine glucose: Abnormal low only | 0 | 0 | 0
  Urine glucose: Abnormal high only | 0 | 0 | 0
  Urine glucose: Abnormal low and abnormal high | 0 | 0 | 0
  Urine ketones: number analyzed (Participants) | 2 | 2 | 4
  Urine ketones: Normal | 1 | 2 | 4
  Urine ketones: Abnormal low only | 0 | 0 | 0
  Urine ketones: Abnormal high only | 1 | 0 | 0
  Urine ketones: Abnormal low and abnormal high | 0 | 0 | 0
  Urine nitrite: number analyzed (Participants) | 2 | 0 | 0
  Urine nitrite: Normal | 2 | 0 | 0
  Urine nitrite: Abnormal low only | 0 | 0 | 0
  Urine nitrite: Abnormal high only | 0 | 0 | 0
  Urine nitrite: Abnormal low and abnormal high | 0 | 0 | 0
  Urine leukocyte esterase: number analyzed (Participants) | 2 | 0 | 0
  Urine leukocyte esterase: Normal | 1 | 0 | 0
  Urine leukocyte esterase: Abnormal low only | 0 | 0 | 0
  Urine leukocyte esterase: Abnormal high only | 1 | 0 | 0
  Urine leukocyte esterase: Abnormal low and abnormal high | 0 | 0 | 0
  Urine erythrocytes: number analyzed (Participants) | 2 | 2 | 4
  Urine erythrocytes: Normal | 2 | 2 | 4
  Urine erythrocytes: Abnormal low only | 0 | 0 | 0
  Urine erythrocytes: Abnormal high only | 0 | 0 | 0
  Urine erythrocytes: Abnormal low and abnormal high | 0 | 0 | 0
  Urine leukocytes: number analyzed (Participants) | 2 | 2 | 4
  Urine leukocytes: Normal | 1 | 1 | 3
  Urine leukocytes: Abnormal low only | 0 | 0 | 0
  Urine leukocytes: Abnormal high only | 1 | 1 | 1
  Urine leukocytes: Abnormal low and abnormal high | 0 | 0 | 0

5. Primary Outcome: Number of Participants With DLTs: Combination Cohort 1
Description: as for outcome 1
Time Frame: Day 1 up to Day 28 of Cycle 1 (28 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Participants | 0

6. Primary Outcome: Number of Participants With TEAEs, Serious TEAEs, Treatment Related TEAEs, Grade 3 or 4 TEAEs Based on NCI CTCAE v4.0: Combination Cohort 1
Description: AE: any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Serious AE: any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. TEAEs: events absent before treatment or that worsened relative to pretreatment state. Treatment-related TEAE: any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to drug was assessed by the Investigator. NCI-CTCAE Grade: Grade 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4= life-threatening consequence, urgent intervention indicated.
Time Frame: Day 1 up to 28 days after last dose of study drug (maximum up to 514 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Participants
  TEAEs | 6
  Serious TEAEs | 1
  Treatment Related TEAEs | 6
  Grade 3 or 4 TEAEs | 4

7. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs Abnormalities: Combination Cohort 1
Description: as for outcome 3
Time Frame: Baseline up to maximum 486 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Participants | 0

8. Primary Outcome: Number of Participants With Worst On-study Laboratory Abnormalities: Combination Cohort 1
Description: Laboratory parameters included- hematology: lymphocytes/leukocytes (%), neutrophils/leukocytes (%), basophils/leukocytes (%), eosinophils/leukocytes (%), monocytes/leukocytes (%), prothrombin time (sec), blasts/leukocytes (%); clinical chemistry: lactate dehydrogenase (u/l), protein (g/l), BUN (mmol/l), urate (mmol/l), chloride (mmol/l), calcium (mmol/l); urinalysis: specific gravity (scalar), pH (scalar), urine glucose (scalar), ketones (scalar), nitrite, leukocyte esterase, urine erythrocytes (scalar), urine leukocytes (scalar). In this outcome measure participants for each laboratory parameter were evaluated as normal, abnormal low only, abnormal high only or abnormal low and an abnormal high. Laboratory values were as per laboratory normal ranges. Values above normal range = abnormal high and below range = abnormal low. Participants with both an abnormal low and an abnormal high value while on study were reported as 'Abnormal low and Abnormal high'.
Time Frame: Baseline up to maximum 514 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Participants
  Lymphocytes/Leukocytes: Normal | 0
  Lymphocytes/Leukocytes: Abnormal low only | 2
  Lymphocytes/Leukocytes: Abnormal high only | 2
  Lymphocytes/Leukocytes: Abnormal low and abnormal high | 2
  Neutrophils/Leukocytes: Normal | 1
  Neutrophils/Leukocytes: Abnormal low only | 4
  Neutrophils/Leukocytes: Abnormal high only | 0
  Neutrophils/Leukocytes: Abnormal low and abnormal high | 1
  Basophils/Leukocytes: Normal | 5
  Basophils/Leukocytes: Abnormal low only | 0
  Basophils/Leukocytes: Abnormal high only | 1
  Basophils/Leukocytes: Abnormal low and abnormal high | 0
  Eosinophils/Leukocytes: Normal | 4
  Eosinophils/Leukocytes: Abnormal low only | 1
  Eosinophils/Leukocytes: Abnormal high only | 1
  Eosinophils/Leukocytes: Abnormal low and abnormal high | 0
  Monocytes/Leukocytes: Normal | 0
  Monocytes/Leukocytes: Abnormal low only | 0
  Monocytes/Leukocytes: Abnormal high only | 4
  Monocytes/Leukocytes: Abnormal low and abnormal high | 2
  Prothrombin time: number analyzed (Participants) | 4
  Prothrombin time: Normal | 1
  Prothrombin time: Abnormal low only | 0
  Prothrombin time: Abnormal high only | 3
  Prothrombin time: Abnormal low and abnormal high | 0
  Blasts/Leukocytes: number analyzed (Participants) | 1
  Blasts/Leukocytes: Normal | 0
  Blasts/Leukocytes: Abnormal low only | 0
  Blasts/Leukocytes: Abnormal high only | 1
  Blasts/Leukocytes: Abnormal low and abnormal high | 0
  Lactate dehydrogenase: Normal | 0
  Lactate dehydrogenase: Abnormal low only | 1
  Lactate dehydrogenase: Abnormal high only | 4
  Lactate dehydrogenase: Abnormal low and abnormal high | 1
  Protein: Normal | 0
  Protein: Abnormal low only | 6
  Protein: Abnormal high only | 0
  Protein: Abnormal low and abnormal high | 0
  BUN: Normal | 3
  BUN: Abnormal low only | 0
  BUN: Abnormal high only | 3
  BUN: Abnormal low and abnormal high | 0
  Urate: Normal | 2
  Urate: Abnormal low only | 3
  Urate: Abnormal high only | 1
  Urate: Abnormal low and abnormal high | 0
  Chloride: Normal | 3
  Chloride: Abnormal low only | 0
  Chloride: Abnormal high only | 3
  Chloride: Abnormal low and abnormal high | 0
  Calcium: Normal | 1
  Calcium: Abnormal low only | 5
  Calcium: Abnormal high only | 0
  Calcium: Abnormal low and abnormal high | 0
  Urine specific gravity: Normal | 6
  Urine specific gravity: Abnormal low only | 0
  Urine specific gravity: Abnormal high only | 0
  Urine specific gravity: Abnormal low and abnormal high | 0
  Urine pH: Normal | 5
  Urine pH: Abnormal low only | 0
  Urine pH: Abnormal high only | 1
  Urine pH: Abnormal low and abnormal high | 0
  Urine glucose: number analyzed (Participants) | 2
  Urine glucose: Normal | 2
  Urine glucose: Abnormal low only | 0
  Urine glucose: Abnormal high only | 0
  Urine glucose: Abnormal low and abnormal high | 0
  Urine ketones: number analyzed (Participants) | 2
  Urine ketones: Normal | 2
  Urine ketones: Abnormal low only | 0
  Urine ketones: Abnormal high only | 0
  Urine ketones: Abnormal low and abnormal high | 0
  Urine nitrite: number analyzed (Participants) | 2
  Urine nitrite: Normal | 2
  Urine nitrite: Abnormal low only | 0
  Urine nitrite: Abnormal high only | 0
  Urine nitrite: Abnormal low and abnormal high | 0
  Urine leukocyte esterase: number analyzed (Participants) | 2
  Urine leukocyte esterase: Normal | 2
  Urine leukocyte esterase: Abnormal low only | 0
  Urine leukocyte esterase: Abnormal high only | 0
  Urine leukocyte esterase: Abnormal low and abnormal high | 0
  Urine erythrocytes: number analyzed (Participants) | 3
  Urine erythrocytes: Normal | 1
  Urine erythrocytes: Abnormal low only | 0
  Urine erythrocytes: Abnormal high only | 2
  Urine erythrocytes: Abnormal low and abnormal high | 0
  Urine leukocytes: number analyzed (Participants) | 3
  Urine leukocytes: Normal | 1
  Urine leukocytes: Abnormal low only | 0
  Urine leukocytes: Abnormal high only | 2
  Urine leukocytes: Abnormal low and abnormal high | 0

9. Primary Outcome: Number of Participants With DLTs: Combination Cohort 2
Description: as for outcome 1
Time Frame: Day -3 up to anytime between Day 21 and Day 28 of first induction cycle (24 to 31 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin: Participants with previously untreated AML/high-risk MDS and fit for intensive chemotherapy, participants started receiving PF-04449913 100 mg tablets QD from Day -3 up to Day 28 for first induction cycle and then continuously QD from Cycle 1/Day 1 in 28 day cycles for rest of treatment duration along with Cytarabine 100 mg/m^2 was administered daily by continuous IV infusion for first 7 days of Cycle and Daunorubicin 60 mg/m^2 daily IV for first 3 days of Cycle. Participants with <= 5% bone marrow blasts had second cycle of induction. Participants achieving a complete response after the completion of induction therapy were eligible to begin consolidation cycles. During consolidation, participants received PF-04449913 100 mg tablets orally QD in 28 day cycle along with Cytarabine 1g/m^2 QD on Day 1, 3 and 5 of 28 day cycle. Consolidation was of 2 to 4 cycles. Post-consolidation participants received PF-04449913 100 mg tablets orally QD in 28-day cycle for maintenance up to maximum of 6 cycles.
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Participants | 1

10. Primary Outcome: Number of Participants With TEAEs, Serious TEAEs, Treatment Related TEAEs, Grade 3 or 4 TEAEs Based on NCI CTCAE v4.0: Combination Cohort 2
Description: as for outcome 6
Time Frame: Day 1 up to 28 days after last dose of study drug (maximum up to 371 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Participants
  TEAEs | 6
  Serious TEAEs | 4
  Treatment Related TEAEs | 6
  Grade 3 or 4 TEAEs | 4

11. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs Abnormalities: Combination Cohort 2
Description: as for outcome 3
Time Frame: Baseline up to maximum 343 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Participants | 0

12. Primary Outcome: Number of Participants With Worst On-study Laboratory Abnormalities: Combination Cohort 2
Description: Laboratory parameters included- hematology: lymphocytes/leukocytes (%), neutrophils/leukocytes (%), basophils/leukocytes (%), eosinophils/leukocytes (%), monocytes/leukocytes (%), prothrombin time (sec), blasts/leukocytes (%); clinical chemistry: lactate dehydrogenase (u/l), protein (g/l), BUN (mmol/l), urate (mmol/l), chloride (mmol/l), calcium (mmol/l); urinalysis: specific gravity (scalar), pH (scalar), urine glucose (scalar), ketones (scalar), urine erythrocytes (scalar), urine leukocytes (scalar). In this outcome measure participants for each laboratory parameter were evaluated as normal, abnormal low only, abnormal high only or abnormal low and an abnormal high. Participants that had both an abnormal low and an abnormal high value while on study were reported as 'Abnormal low and Abnormal high'.
Time Frame: Baseline up to maximum 371 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication. Here "number of participants analyzed" signifies participants evaluable for the specific parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Participants
  Lymphocytes/Leukocytes: Normal | 0
  Lymphocytes/Leukocytes: Abnormal low only | 0
  Lymphocytes/Leukocytes: Abnormal high only | 0
  Lymphocytes/Leukocytes: Abnormal low and abnormal high | 6
  Neutrophils/Leukocytes: Normal | 0
  Neutrophils/Leukocytes: Abnormal low only | 1
  Neutrophils/Leukocytes: Abnormal high only | 0
  Neutrophils/Leukocytes: Abnormal low and abnormal high | 5
  Basophils/Leukocytes: Normal | 4
  Basophils/Leukocytes: Abnormal low only | 1
  Basophils/Leukocytes: Abnormal high only | 1
  Basophils/Leukocytes: Abnormal low and abnormal high | 0
  Eosinophils/Leukocytes: Normal | 1
  Eosinophils/Leukocytes: Abnormal low only | 2
  Eosinophils/Leukocytes: Abnormal high only | 1
  Eosinophils/Leukocytes: Abnormal low and abnormal high | 2
  Monocytes/Leukocytes: Normal | 0
  Monocytes/Leukocytes: Abnormal low only | 0
  Monocytes/Leukocytes: Abnormal high only | 2
  Monocytes/Leukocytes: Abnormal low and abnormal high | 4
  Prothrombin time: Normal | 1
  Prothrombin time: Abnormal low only | 0
  Prothrombin time: Abnormal high only | 5
  Prothrombin time: Abnormal low and abnormal high | 0
  Blasts/Leukocytes: number analyzed (Participants) | 4
  Blasts/Leukocytes: Normal | 0
  Blasts/Leukocytes: Abnormal low only | 0
  Blasts/Leukocytes: Abnormal high only | 4
  Blasts/Leukocytes: Abnormal low and abnormal high | 0
  Lactate dehydrogenase: Normal | 2
  Lactate dehydrogenase: Abnormal low only | 0
  Lactate dehydrogenase: Abnormal high only | 4
  Lactate dehydrogenase: Abnormal low and abnormal high | 0
  Protein: Normal | 0
  Protein: Abnormal low only | 6
  Protein: Abnormal high only | 0
  Protein: Abnormal low and abnormal high | 0
  BUN: Normal | 1
  BUN: Abnormal low only | 2
  BUN: Abnormal high only | 3
  BUN: Abnormal low and abnormal high | 0
  Urate: Normal | 0
  Urate: Abnormal low only | 5
  Urate: Abnormal high only | 0
  Urate: Abnormal low and abnormal high | 1
  Chloride: Normal | 3
  Chloride: Abnormal low only | 3
  Chloride: Abnormal high only | 0
  Chloride: Abnormal low and abnormal high | 0
  Calcium: Normal | 0
  Calcium: Abnormal low only | 5
  Calcium: Abnormal high only | 0
  Calcium: Abnormal low and abnormal high | 1
  Urine specific gravity: Normal | 3
  Urine specific gravity: Abnormal low only | 2
  Urine specific gravity: Abnormal high only | 1
  Urine specific gravity: Abnormal low and abnormal high | 0
  Urine pH: Normal | 5
  Urine pH: Abnormal low only | 0
  Urine pH: Abnormal high only | 1
  Urine pH: Abnormal low and abnormal high | 0
  Urine glucose: number analyzed (Participants) | 1
  Urine glucose: Normal | 1
  Urine glucose: Abnormal low only | 0
  Urine glucose: Abnormal high only | 0
  Urine glucose: Abnormal low and abnormal high | 0
  Urine ketones: number analyzed (Participants) | 1
  Urine ketones: Normal | 1
  Urine ketones: Abnormal low only | 0
  Urine ketones: Abnormal high only | 0
  Urine ketones: Abnormal low and abnormal high | 0
  Urine erythrocytes: number analyzed (Participants) | 1
  Urine erythrocytes: Normal | 1
  Urine erythrocytes: Abnormal low only | 0
  Urine erythrocytes: Abnormal high only | 0
  Urine erythrocytes: Abnormal low and abnormal high | 0
  Urine leukocytes: number analyzed (Participants) | 1
  Urine leukocytes: Normal | 1
  Urine leukocytes: Abnormal low only | 0
  Urine leukocytes: Abnormal high only | 0
  Urine leukocytes: Abnormal low and abnormal high | 0

13. Primary Outcome: Percentage of Participants Achieving Disease Modifying Response (DMR): Expansion Cohort
Description: DMR included complete remission (CR), CR with incomplete blood count recovery (Cri), morphologic leukemia-free state (MLFS), marrow CR (mCR) and partial remission (PR). CR: >=11 gram per deciliter (g/dL) hemoglobin (Hgb), >=1*10^9 neutrophils (L), >=100*10^9 platelets (L), 0% blasts, <=5% bone marrow blasts (BMB), normal maturation of all cell lines, if had persistent dysplasia. . CRi: <1000 neutrophils (mcL), <100000 platelets (mcL), <5% BMB, either neutrophils or platelets not recovered, no extramedullary disease (EMD). MLFS: 1000 neutrophils (mcL) and <100000 platelets (mcL), <5% BMB, neutrophils and platelets not recovered, flow cytometry negative, no EMD. PR: >=1000 neutrophils (mcL), >=100000 platelets (mcL), decrease to 5-25 and >=50% decrease from start, Blasts <=5% if Auer rod positive. mCR: hematologic improvement (HI) response, <=5% and decreased by >=50% BMB. PR: decrease by >=50% but still >5% BMB.
Time Frame: Baseline up to maximum 736 days
Population: Full analysis set (FAS) included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 15
Percentage of participants | 46.7 [24.4 to 70.0]
Statistical Analysis 1: Comparison: Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg; Test type: Other; p < .0001, Exact test for a single proportion — An exact test for a single proportion (1-sided significance level: 0.05) was used

14. Primary Outcome: Number of Participants With DLTs: Combination Cohort 3
Description: as for outcome 1
Time Frame: Day 1 up to Day 28 of Cycle 1 (28 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Participants | 0

15. Primary Outcome: Number of Participants With TEAEs, Serious TEAEs, Treatment Related TEAEs, Grade 3 or 4 TEAEs Based on NCI CTCAE v4.0: Combination Cohort 3
Description: as for outcome 6
Time Frame: Day 1 up to 28 days after last dose of study drug (maximum up to 869 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Participants
  TEAEs | 6
  Serious TEAEs | 1
  Treatment related TEAEs | 6
  Grade 3 or 4 TEAEs | 5

16. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs Abnormalities: Combination Cohort 3
Description: as for outcome 3
Time Frame: Baseline up to maximum 841 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Participants | 0

17. Primary Outcome: Number of Participants With Worst On-study Laboratory Abnormalities: Combination Cohort 3
Description: Laboratory parameters included- hematology: lymphocytes/leukocytes (%), neutrophils/leukocytes (%), basophils/leukocytes (%), eosinophils/leukocytes (%), monocytes/leukocytes (%), blasts/leukocytes (%); clinical chemistry: lactate dehydrogenase (u/l), protein (g/l), BUN (mmol/l), urate (mmol/l), chloride (mmol/l), calcium (mmol/l); urinalysis: specific gravity (scalar), pH (scalar), urine glucose (scalar), ketones (scalar), nitrite, leukocyte esterase, urine erythrocytes (scalar), urine leukocytes (scalar). In this outcome measure participants for each laboratory parameter were evaluated as normal, abnormal low only, abnormal high only or abnormal low and an abnormal high. Participants that had both an abnormal low and an abnormal high value while on study were reported as 'Abnormal low and Abnormal high'.
Time Frame: Baseline up to maximum 869 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Participants
  Lymphocytes/Leukocytes: Normal | 0
  Lymphocytes/Leukocytes: Abnormal low only | 2
  Lymphocytes/Leukocytes: Abnormal high only | 1
  Lymphocytes/Leukocytes: Abnormal low and abnormal high | 3
  Neutrophils/Leukocytes: Normal | 0
  Neutrophils/Leukocytes: Abnormal low only | 5
  Neutrophils/Leukocytes: Abnormal high only | 0
  Neutrophils/Leukocytes: Abnormal low and abnormal high | 1
  Basophils/Leukocytes: Normal | 4
  Basophils/Leukocytes: Abnormal low only | 0
  Basophils/Leukocytes: Abnormal high only | 1
  Basophils/Leukocytes: Abnormal low and abnormal high | 1
  Eosinophils/Leukocytes: Normal | 3
  Eosinophils/Leukocytes: Abnormal low only | 1
  Eosinophils/Leukocytes: Abnormal high only | 0
  Eosinophils/Leukocytes: Abnormal low and abnormal high | 2
  Monocytes/Leukocytes: Normal | 0
  Monocytes/Leukocytes: Abnormal low only | 2
  Monocytes/Leukocytes: Abnormal high only | 3
  Monocytes/Leukocytes: Abnormal low and abnormal high | 1
  Blasts/Leukocytes: number analyzed (Participants) | 2
  Blasts/Leukocytes: Normal | 0
  Blasts/Leukocytes: Abnormal low only | 0
  Blasts/Leukocytes: Abnormal high only | 2
  Blasts/Leukocytes: Abnormal low and abnormal high | 0
  Lactate dehydrogenase: Normal | 0
  Lactate dehydrogenase: Abnormal low only | 1
  Lactate dehydrogenase: Abnormal high only | 4
  Lactate dehydrogenase: Abnormal low and abnormal high | 1
  Protein: Normal | 2
  Protein: Abnormal low only | 4
  Protein: Abnormal high only | 0
  Protein: Abnormal low and abnormal high | 0
  BUN: Normal | 3
  BUN: Abnormal low only | 0
  BUN: Abnormal high only | 2
  BUN: Abnormal low and abnormal high | 1
  Urate: Normal | 2
  Urate: Abnormal low only | 2
  Urate: Abnormal high only | 1
  Urate: Abnormal low and abnormal high | 1
  Chloride: Normal | 2
  Chloride: Abnormal low only | 4
  Chloride: Abnormal high only | 0
  Chloride: Abnormal low and abnormal high | 0
  Calcium: Normal | 0
  Calcium: Abnormal low only | 6
  Calcium: Abnormal high only | 0
  Calcium: Abnormal low and abnormal high | 0
  Urine specific gravity: Normal | 5
  Urine specific gravity: Abnormal low only | 0
  Urine specific gravity: Abnormal high only | 1
  Urine specific gravity: Abnormal low and abnormal high | 0
  Urine pH: Normal | 5
  Urine pH: Abnormal low only | 0
  Urine pH: Abnormal high only | 1
  Urine pH: Abnormal low and abnormal high | 0
  Urine glucose: number analyzed (Participants) | 2
  Urine glucose: Normal | 2
  Urine glucose: Abnormal low only | 0
  Urine glucose: Abnormal high only | 0
  Urine glucose: Abnormal low and abnormal high | 0
  Urine ketones: number analyzed (Participants) | 2
  Urine ketones: Normal | 2
  Urine ketones: Abnormal low only | 0
  Urine ketones: Abnormal high only | 0
  Urine ketones: Abnormal low and abnormal high | 0
  Urine nitrite: number analyzed (Participants) | 2
  Urine nitrite: Normal | 2
  Urine nitrite: Abnormal low only | 0
  Urine nitrite: Abnormal high only | 0
  Urine nitrite: Abnormal low and abnormal high | 0
  Urine leukocyte esterase: number analyzed (Participants) | 2
  Urine leukocyte esterase: Normal | 2
  Urine leukocyte esterase: Abnormal low only | 0
  Urine leukocyte esterase: Abnormal high only | 0
  Urine leukocyte esterase: Abnormal low and abnormal high | 0
  Urine erythrocytes: number analyzed (Participants) | 2
  Urine erythrocytes: Normal | 2
  Urine erythrocytes: Abnormal low only | 0
  Urine erythrocytes: Abnormal high only | 0
  Urine erythrocytes: Abnormal low and abnormal high | 0
  Urine leukocytes: number analyzed (Participants) | 2
  Urine leukocytes: Normal | 2
  Urine leukocytes: Abnormal low only | 0
  Urine leukocytes: Abnormal high only | 0
  Urine leukocytes: Abnormal low and abnormal high | 0

18. Secondary Outcome: Single Dose- Maximum Observed Plasma Concentration (Cmax) of PF-04449913: Monotherapy Cohort
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 24, 48, 72 hours post PF-04449913 dosing on Day -5 of Cycle 1
Population: Pharmacokinetic (PK) parameter analysis set included all treated participants with at least 1 PK parameters of interest of any of the study drugs.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
nanogram per milliliter | 281.5 (96) | 321.1 (57) | 1019 (25)

19. Secondary Outcome: Single Dose- Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04449913: Monotherapy Cohort
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 24, 48, 72 hours post PF-04449913 dosing on Day -5 of Cycle 1
Population: PK parameter analysis set included all treated participants with at least 1 PK parameters of interest of any of the study drugs.
Measure: Median (Full Range); unit: Hours
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Hours | 1.970 [1.08 to 4.00] | 3.955 [2.02 to 7.28] | 1.950 [0.933 to 4.03]

20. Secondary Outcome: Single Dose- Terminal Plasma Half-life (T1/2) of PF-04449913: Monotherapy Cohort
Description: Terminal plasma half-life is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 24, 48, 72 hours post PF-04449913 dosing on Day -5 of Cycle 1
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Hours | 17.83 (1.0214) | 30.70 (5.7498) | 18.67 (3.5359)

21. Secondary Outcome: Single Dose- Area Under the Plasma Concentration Curve: From Time Zero to End of Dosing Interval (AUCtau), From Time Zero to Last Quantifiable Concentration (AUClast) and From Time Zero to Infinity (AUCinf) of PF-04449913 for Monotherapy Cohort
Description: AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours. AUClast = area under the curve from time zero to last quantifiable concentration. AUCinf = AUClast + (Clast/kel), where Clast = predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and where kel = terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: AUCtau: 0 to 24, 24 to 48, 48 to 72 hours post PF-04449913 dosing on Day -5 of Cycle 1; AUClast and AUCinf: Pre-dose and 0.5, 1, 2, 4, 8, 24, 48, 72 hours post PF-04449913 dosing on Day -5 of Cycle 1
Population: PK parameter analysis set included all treated participants with at least 1 PK parameter of interest of any of the study drugs.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Nanogram*hour per milliliter
  AUCtau | 2413 (73) | 4499 (51) | 8843 (19)
  AUClast | 3255 (70) | 8911 (63) | 12750 (21)
  AUCinf | 3374 (68) | 9596 (65) | 13160 (20)

22. Secondary Outcome: Single Dose- Clearance (CL/F) of PF-04449913: Monotherapy Cohort
Description: CL/F was defined as apparent total clearance of the drug from plasma after oral administration. CL/F of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 24, 48, 72 hours post PF-04449913 dosing on Day -5 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Liter per hour | 7.415 (68) | 5.210 (65) | 7.599 (20)

23. Secondary Outcome: Single Dose- Volume of Distribution (Vz/F) of PF-04449913: Monotherapy Cohort
Description: Vz/F was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 24, 48, 72 hours post PF-04449913 dosing on Day -5 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Liter | 190.5 (62) | 227.8 (49) | 201.5 (20)

24. Secondary Outcome: Multiple Dose Cmax, Minimum Observed Plasma Concentration (Cmin), Average Observed Plasma Concentration (Cavg), Trough Plasma Concentration (Ctrough) of PF-04449913: Monotherapy Cohort
Description: Cmax = Maximum plasma concentration, observed directly from data. Cmin = Minimum plasma concentration observed directly from data. Cavg = Average plasma concentration over the dosing interval, dosing interval was of 24 hours. Ctrough = Pre-dose concentration, observed directly from data.
Time Frame: Cmax, Cmin: Pre-dose and 0.5, 1, 2, 4, 8, and 24 hours post PF-04449913 dosing on Day 21 of Cycle 1; Cavg: 0 to 24, 24 to 48, 48 to 72 hours post PF-04449913 dosing on Day 21 of Cycle 1; Ctrough: Pre-dose on Day 21 of Cycle 1
Population: PK parameter analysis set included all treated participants with at least 1 PK parameters of interest of any of the study drugs. Here "number of participants analyzed" signifies participants evaluable for the specific parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Nanogram per milliliter
  Cmax: number analyzed (Participants) | 3 | 3 | 6
  Cmax | 356.9 (90) | 542.2 (10) | 1330 (12)
  Cmin: number analyzed (Participants) | 3 | 3 | 6
  Cmin | 84.94 (127) | 237.2 (36) | 333.9 (34)
  Cavg: number analyzed (Participants) | 3 | 3 | 6
  Cavg | 190.5 (99) | 388.1 (14) | 645.8 (26)
  Ctrough: number analyzed (Participants) | 3 | 3 | 6
  Ctrough | 87.87 (139) | 240.0 (37) | 342.9 (35)

25. Secondary Outcome: Multiple Dose- Tmax of PF-04449913: Monotherapy Cohort
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, and 24 hours post PF-04449913 dosing on Day 21 of Cycle 1
Population: PK parameter analysis set included all treated participants with at least 1 PK parameters of interest of any of the study drugs. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Hours
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 3 | 6
Hours | 3.970 [3.90 to 4.02] | 4.000 [3.93 to 7.25] | 1.950 [0.933 to 3.90]

26. Secondary Outcome: Multiple Dose- AUCtau of PF-04449913: Monotherapy Cohort
Description: as for outcome 21
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, and 24 hours post PF-04449913 dosing Day 21 of Cycle 1
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 3 | 6
Nanogram*hour per milliliter | 4561 (99) | 9299 (14) | 15480 (26)

27. Secondary Outcome: Multiple Dose- Clearance (CL/F) of PF-04449913: Monotherapy Cohort
Description: as for outcome 22
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, and 24 hours post PF-04449913 dosing Day 21 of Cycle 1
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 3 | 6
Liter per hour | 5.467 (98) | 5.369 (14) | 6.452 (25)

28. Secondary Outcome: Multiple Dose- Accumulation Ratio (Rac) of PF-04449913: Monotherapy Cohort
Description: Rac was the observed accumulation ratio for AUCtau, determined as ratio of Day 21 AUCtau to Day -5 AUCtau. AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours.
Time Frame: 0 to 24, 24 to 48, 48 to 72 hours post PF-04449913 dosing on Day -5 and Day 21 of Cycle 1
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 3 | 6
Ratio | 1.893 (40) | 2.076 (67) | 1.752 (25)

29. Secondary Outcome: Multiple Dose- Steady State Accumulation Ratio (Rss) of PF-04449913: Monotherapy Cohort
Description: Rss = Ratio of Day 21 AUCtau to Day -5 AUCinf. AUCinf = AUClast + (Clast/kel), where Clast = predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and where kel = terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours.
Time Frame: AUCtau: 0 to 24, 24 to 48, 48 to 72 hours post PF-04449913 dosing on Day 21 of Cycle 1; AUCinf: Pre-dose and 0.5, 1, 2, 4, 8, 24, 48, 72 hours post PF-04449913 dosing on Day -5 of Cycle 1
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 3 | 6
Ratio | 1.355 (32) | 1.017 (85) | 1.176 (18)

30. Secondary Outcome: Ratio of GLI1 Levels at Baseline to Day 21 Cycle 1: Monotherapy Cohort
Description: Biomarker assessments were used to understand the in vivo mechanism of action of PF-04449913, as well as potential mechanisms of resistance. In this outcome measure ratio of GLI1 levels (mRNA, fresh tissue) at baseline to day 21 cycle 1 is reported.
Time Frame: Baseline, Day 21 of Cycle 1 (Unspecified- at any time on Day 21)
Population: The PD analysis set included all enrolled participants who received at least 1 dose of PF-04449913 and had at least 1 pharmacodynamic parameter in active treatment period. Here "number of participants analyzed" signifies participants evaluable for the specific parameter.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 2 | 3 | 5
Ratio | 1.170 (0.2769) | 1.588 (0.1773) | 1.695 (0.1108)

31. Secondary Outcome: Number of Participants With Best Response: Monotherapy Cohort
Description: Best response observed for: CR, Cri, MLFS, PR, PRi, CytogeneticCR(CRc), MolecularCR(CRm). For AML-CR:neutrophils(nt) [mcL]>=1000, platelets(pt)[mcL]>=10^5, BMB<5%. CRi:nt(mcL)<1000/pt(mcL)<10^5, BMB<5%. MLFS:nt(mcL)1000 and pt(mcL)<10^5, BMB<5%. PR:nt(mcL)>=1000, pt(mcL)>=10^5, decrease to 5-25 and >=50% decrease from start. PRi: nt<1000, <10^5. CRc: nt(mcL)>1,000, pt(mcL)>10^5, BMB<5%. CRm: nt(mcL)>1,000, pt(uL)>10^5, BMB<5%. For myelodysplasia-CR: hemoglobin(Hgb)[gram per deciliter{g/dL}]>=11, nt(L)>=1*10^9, pt(L)>=100*10^9, blasts0%, BMB<=5%. mCR:<=5% and decreased by >=50% BMB. PR:decrease by>=50% with >5% BMB, CRc: disappearance of chromosomal abnormality, no new appearance, PRc:>=50% reduced chromosomal abnormality. For myleofibrosis-CR: hgb(g/L)>=110, nt(L)>=1*10^9, pt(L)>=100*10^9, All <=ULN, BMB <=5%. PR: hgb>=110, nt(L)>=1*10^9, pt(L)>=100*10^9. CML- PR: 1-35% Philadelphia chromosome(PC) positive(+) cells, CR:0% PC+ cells. Responses with at least 1 participant were reported.
Time Frame: Day 1 up to End of Treatment (25 mg: maximum up to 108 days; 50 mg: maximum up to 151 days; 100 mg: maximum up to 444 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1. Here, "number of participants analyzed" signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Cohort: PF-04449913 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg
Number analyzed (Participants) | 3 | 4 | 6
Participants
  Morphologic CR: AML: number analyzed (Participants) | 1 | 2 | 4
  Morphologic CR: AML | 0 | 0 | 1
  Morphologic CRi: AML: number analyzed (Participants) | 1 | 2 | 4
  Morphologic CRi: AML | 0 | 0 | 1
  MLFs: AML: number analyzed (Participants) | 1 | 2 | 4
  MLFs: AML | 0 | 0 | 1
  Stable disease: AML: number analyzed (Participants) | 1 | 2 | 4
  Stable disease: AML | 1 | 1 | 2
  Treatment failure: AML: number analyzed (Participants) | 1 | 2 | 4
  Treatment failure: AML | 1 | 1 | 3
  Marrow complete remission: MDS | 0 | 0 | 1
  Stable disease: MDS: number analyzed (Participants) | 2 | 1 | 1
  Stable disease: MDS | 1 | 1 | 1
  Disease progression: MDS: number analyzed (Participants) | 2 | 1 | 1
  Disease progression: MDS | 0 | 1 | 0
  Treatment failure: MDS: number analyzed (Participants) | 2 | 1 | 1
  Treatment failure: MDS | 1 | 0 | 0
  Stable disease: CML: number analyzed (Participants) | 0 | 1 | 6
  Stable disease: CML | 0 | 1 | 0
  Disease progression: CML: number analyzed (Participants) | 0 | 1 | 0
  Disease progression: CML | 0 | 1 | 0

32. Secondary Outcome: Multiple Dose- Cmax, Cmin, Cavg, and Ctrough of PF-04449913: Combination Cohort 1
Description: as for outcome 24
Time Frame: Cmax, Cmin: Pre-dose and 0.5, 1, 2, 4, 6 and 24 hours post PF-04449913 dose on Day 10 and 21 of Cycle 1; Cavg: 0 to 24 hours post PF-04449913 dose on Day 10 and 21 of Cycle; Ctrough: Pre-dose on Day 10 and 21 of Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Nanogram per milliliter
  Cmax: Cycle 1/Day 10 | 1172 (38)
  Cmin: Cycle 1/Day 10 | 317.6 (91)
  Cavg: Cycle 1/Day 10 | 648.3 (58)
  Ctrough: Cycle 1/Day 10 | 330.7 (92)
  Cmax: Cycle 1/Day 21 | 1317 (86)
  Cmin: Cycle 1/Day 21 | 341.6 (172)
  Cavg: Cycle 1/Day 21 | 670.5 (113)
  Ctrough: Cycle 1/Day 21 | 376.2 (142)

33. Secondary Outcome: Multiple Dose- Tmax of PF-04449913: Combination Cohort 1
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6 and 24 hours post PF-04449913 dose on Day 10 and Day 21 of Cycle 1
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Hours
  Cycle 1/Day 10 | 3.950 [1.00 to 4.05]
  Cycle 1/Day 21 | 1.935 [0.967 to 2.00]

34. Secondary Outcome: Multiple Dose- AUCtau of PF-04449913: Combination Cohort 1
Description: AUCtau was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours.
Time Frame: 0 to 24 hours post PF-04449913 dose on Day 10 and Day 21 of Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Nanogram*hour per milliliter
  Cycle 1/Day 10 | 15560 (58)
  Cycle 1/Day 21 | 16070 (113)

35. Secondary Outcome: Multiple Dose- CL/F of PF-04449913: Combination Cohort 1
Description: as for outcome 22
Time Frame: Pre-dose and 0.5, 1, 2, 4, 6 and 24 hours post PF-04449913 dose on Day 10 and Day 21 of Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Liter per hour
  Cycle 1/Day 10 | 6.428 (58)
  Cycle 1/Day 21 | 6.223 (113)

36. Secondary Outcome: Multiple Dose- Cmax, Cmin, Cavg, and Ctrough of Cytarabine: Combination Cohort 1
Description: LDAC= low dose ara-cytarabine/low dose cytarabine. Cmax = Maximum plasma concentration, observed directly from data. Cmin = Minimum plasma concentration observed directly from data. Cavg = Average plasma concentration over the dosing interval, dosing interval was of 24 hours, dosing interval was of 12 hours. Ctrough = Pre-dose concentration, observed directly from data.
Time Frame: Cmax, Cmin: Pre-dose and 0.25, 0.5, 1, 2, 4 and 6 hours post LDAC dosing on Day 2 and Day 10 of Cycle 1; Cavg: 0 to 12 hours post LDAC dosing on Day 2 and Day 10 of Cycle 1; Ctrough: Pre-LDAC dose on Day 2 and Day 10 of Cycle 1
Population: PK parameter analysis set included all treated participants with at least 1 PK parameters of interest of any of the study drugs. Here, "number of participants analyzed" signifies participants evaluable for the specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Nanogram per milliliter
  Cmax: Cycle 1/Day 2 | 82.88 (105)
  Cmin: Cycle 1/Day 2 | NA (NA) — Cmin was not estimable as the analyte was not detected for any participant.
  Cavg: Cycle 1/Day 2 | 6.511 (82)
  Ctrough: Cycle 1/Day 2 | NA (NA) — Ctrough was not estimable as the analyte was not detected for any participant.
  Cmax: Cycle 1/Day 10 | 106.7 (29)
  Cmin: Cycle 1/Day 10 | 0.5903 (11)
  Cavg: Cycle 1/Day 10: number analyzed (Participants) | 5
  Cavg: Cycle 1/Day 10 | 8.135 (18)
  Ctrough: Cycle 1/Day 10 | 0.5903 (11)

37. Secondary Outcome: Multiple Dose- Tmax of Cytarabine: Combination Cohort 1
Description: LDAC= low dose ara-cytarabine/low dose cytarabine.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4 and 6 hours post LDAC dosing on Day 2 and Day 10 of Cycle 1
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Hours
  Cycle 1/Day 2 | 0.2500 [0.233 to 0.250]
  Cycle 1/Day 10 | 0.2500 [0.233 to 0.317]

38. Secondary Outcome: Multiple Dose- T1/2 of Cytarabine: Combination Cohort 1
Description: LDAC= low dose ara-cytarabine/low dose cytarabine. Terminal plasma half-life is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4 and 6 hours post LDAC dosing on Day 2 and Day 10 of Cycle 1
Population: PK parameter analysis set included all treated participants with at least 1 PK parameters of interest of any of the study drugs. Here, "number of participants analyzed" signifies participants evaluable for the specific parameter.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Hours
  Cycle 1/Day 2 | 1.027 (0.27844)
  Cycle 1/Day 10: number analyzed (Participants) | 5
  Cycle 1/Day 10 | 0.8618 (0.029677)

39. Secondary Outcome: Multiple Dose- AUCinf and AUCtau of Cytarabine: Combination Cohort 1
Description: LDAC= low dose ara-cytarabine/low dose cytarabine. AUCinf = AUClast + (Clast/kel), where Clast = predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and where kel = terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 12 hours.
Time Frame: AUCinf: Pre-dose and 0.25, 0.5, 1, 2, 4 and 6 hours post LDAC dosing on Day 2 and Day 10 of Cycle 1; AUCtau: 0 to 12 hours post LDAC dosing on Day 2 and Day 10 of Cycle
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Nanogram*hour per milliliter
  AUCinf: Cycle 1/Day 2 | 78.37 (80)
  AUCtau: Cycle 1/Day 2 | 77.97 (82)
  AUCinf: Cycle 1/Day 10: number analyzed (Participants) | 5
  AUCinf: Cycle 1/Day 10 | 97.34 (18)
  AUCtau: Cycle 1/Day 10: number analyzed (Participants) | 5
  AUCtau: Cycle 1/Day 10 | 97.58 (18)

40. Secondary Outcome: Multiple Dose- Cmax, Cmin, and Ctrough of Ara-uridine: Combination Cohort 1
Description: Ara-uridine was a metabolite of cytarabine. Cmax = Maximum plasma concentration, observed directly from data. Cmin = Minimum plasma concentration observed directly from data. Cavg = Average plasma concentration over the dosing interval, dosing interval was of 12 hours. Ctrough = Pre-dose concentration, observed directly from data. Ara-uridine was a metabolite of cytarabine.
Time Frame: Cmax, Cmin: Pre-dose and 0.25, 0.5, 1, 2, 4 and 6 hours post LDAC dosing on Day 2 and Day 10 of Cycle 1; Cavg: 0 to 12 hours post LDAC dosing on Day 2 and Day 10 of Cycle 1; Ctrough: Pre-LDAC dosing on Day 2 and Day 10 of Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Nanogram per milliliter
  Cmax: Cycle 1/Day 2 | 371.6 (37)
  Cmin: Cycle 1/Day 2 | 141.9 (61)
  Ctrough: Cycle 1/Day 2 | 141.9 (61)
  Cmax: Cycle 1/Day 10 | 454.3 (33)
  Cmin: Cycle 1/Day 10 | 201.7 (61)
  Ctrough: Cycle 1/Day 10 | 201.7 (61)

41. Secondary Outcome: Multiple Dose- Tmax of Ara-uridine: Combination Cohort 1
Description: Ara-uridine was a metabolite of cytarabine.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4 and 6 hours post LDAC dosing on Day 2 and Day 10 of Cycle 1
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Hours
  Cycle 1/Day 2 | 1.515 [0.917 to 4.00]
  Cycle 1/Day 10 | 2.000 [1.92 to 4.05]

42. Secondary Outcome: Multiple Dose- Cmax, Cmin, Cavg, and Ctrough of PF-04449913: Combination Cohort 2
Description: as for outcome 24
Time Frame: Cmax, Cmin: Pre-dose, 0.5, 1, 6, and 24 hrs post dose on Day 3, 10 of induction Cycle (IC) 1 and 4 hrs post dose on Day 10 of IC 1; Cavg: 0 to 24 hrs post dose on Day 3 and Day 10 of IC 1; Ctrough: Pre dose on Day 3 and Day 10 of IC 1 (PF-04449913 Dose)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Nanogram per milliliter
  Cmax: Cycle 1/Day 3 | 1047 (40)
  Cmin: Cycle 1/Day 3 | 318.2 (53)
  Cavg: Cycle 1/Day 3 | 650.9 (46)
  Ctrough: Cycle 1/Day 3 | 354.0 (47)
  Cmax: Cycle 1/Day 10 | 1181 (54)
  Cmin: Cycle 1/Day 10 | 356.1 (85)
  Cavg: Cycle 1/Day 10 | 755.2 (58)
  Ctrough: Cycle 1/Day 10 | 359.5 (85)

43. Secondary Outcome: Multiple Dose- Tmax of PF-04449913: Combination Cohort 2
Time Frame: Pre-dose, 0.5, 1, 6, and 24 hours post PF-04449913 dosing on Day 3 of Induction Cycle 1 and pre-dose, 0.5, 1, 4, 6, and 24 hours post PF-04449913 dosing on Day 10 of Induction Cycle 1
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Hours
  Cycle 1/Day 3 | 5.950 [1.00 to 6.13]
  Cycle 1/Day 10 | 5.065 [3.98 to 6.03]

44. Secondary Outcome: Multiple Dose- AUCtau of PF-04449913: Combination Cohort 2
Description: AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours.
Time Frame: as for outcome 43
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Nanogram*hour per milliliter
  Cycle 1/Day 3 | 15630 (46)
  Cycle 1/Day 10 | 18120 (58)

45. Secondary Outcome: Multiple Dose- CL/F of PF-04449913: Combination Cohort 2
Description: as for outcome 22
Time Frame: as for outcome 43
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Liter per hour
  Cycle 1/Day 3 | 6.401 (46)
  Cycle 1/Day 10 | 5.523 (58)

46. Secondary Outcome: Multiple Dose- Cmax, Cmin, Cavg, and Ctrough of Daunorubicin: Combination Cohort 2
Description: as for outcome 24
Time Frame: Cmax, Cmin: Pre-dose, 0.25 (mid-infusion), 0.5 (immediately prior to end of infusion), 1, 4, 6, 24 hours post daunorubicin dosing on Day 3 of induction Cycle (IC) 1; Cavg: 0 to 24 hours post dose on Day 3 of IC 1; Ctrough: Pre-dose on Day 3 of IC 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Nanogram per milliliter
  Cmax | 942.8 (35)
  Cmin | 2.589 (25)
  Cavg | 30.89 (27)
  Ctrough | 2.673 (24)

47. Secondary Outcome: Multiple Dose- Tmax of Daunorubicin: Combination Cohort 2
Time Frame: Pre-dose, 0.25 (mid-infusion), 0.5 (immediately prior to end of infusion), 1, 4, 6, 24 hours post daunorubicin dosing on Day 3 of induction Cycle 1
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Hours | 0.3585 [0.250 to 0.500]

48. Secondary Outcome: Multiple Dose- T1/2 of Daunorubicin: Combination Cohort 2
Description: as for outcome 20
Time Frame: Pre-dose, 0.25 (mid-infusion), 0.5 (immediately prior to end of infusion), 1, 4, 6, 24 hours post daunorubicin dosing on Day 3 of at induction Cycle 1
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Hours | 7.297 (0.65525)

49. Secondary Outcome: Multiple Dose- AUCinf and AUCtau of Daunorubicin: Combination Cohort 2
Description: AUCinf = AUClast + (Clast/kel), where Clast = predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and where kel = terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours.
Time Frame: AUCinf: Pre-dose, 0.25 (mid-infusion), 0.5 (immediately prior to end of infusion), 1, 4, 6, 24 hours post daunorubicin dosing on Day 3 of induction Cycle 1; AUCtau: 0 to 24 hours post daunorubicin dosing on Day 3 of induction Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Nanogram*hour per milliliter
  AUCinf | 770.4 (27)
  AUCtau | 741.6 (27)

50. Secondary Outcome: Multiple Dose- Cmax, Cmin, Cavg, and Ctrough of Daunorubicinol: Combination Cohort 2
Description: Cmax = Maximum plasma concentration, observed directly from data. Cmin = Minimum plasma concentration observed directly from data. Cavg = Average plasma concentration over the dosing interval of 24 hours. Ctrough = Pre-dose concentration, observed directly from data. Daunorubicinol was a metabolite of daunorubicin.
Time Frame: as for outcome 46
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Nanogram per milliliter
  Cmax | 244.4 (37)
  Cmin | 66.38 (21)
  Cavg | 116.7 (13)
  Ctrough | 66.53 (21)

51. Secondary Outcome: Multiple Dose- Tmax of Daunorubicinol: Combination Cohort 2
Description: Daunorubicinol was a metabolite of daunorubicin.
Time Frame: as for outcome 47
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Hours | 0.3585 [0.250 to 0.500]

52. Secondary Outcome: Multiple Dose- AUCtau of Daunorubicinol: Combination Cohort 2
Description: Daunorubicinol was a metabolite of daunorubicin. AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours.
Time Frame: 0 to 24 hours post daunorubicin dosing on Day 3 of induction Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Nanogram*hour per milliliter | 2800 (13)

53. Secondary Outcome: Ratio of GLI1 Levels at Baseline to Day 21 Cycle 1: Combination Cohort 1
Description: as for outcome 30
Time Frame: Baseline, Day 21 of Cycle 1 (Unspecified- at any time on Day 21)
Population: The PD analysis set included all enrolled participants who received at least 1 dose of PF-04449913 and had at least 1 pharmacodynamic parameter in active treatment period. Here, "number of participants analyzed" signifies participants evaluable for the specific parameter.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 5
Ratio | 1.835 (0.3597)

54. Secondary Outcome: Ratio of GLI1 Levels at Baseline to Day 21 Cycle1: Combination Cohort 2
Description: as for outcome 30
Time Frame: Baseline, Day 21 of Cycle 1 (Unspecified- at any time on Day 21)
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 4
Ratio | 1.666 (0.0797)

55. Secondary Outcome: Number of Participants With Best Response: Combination Cohort 1
Description: Best response observed for: CR, Cri, MLFS, PR, PRi, CRc, CRm. Response criteria for participants with AML- CR: neutrophils [mcL] >=1000, platelets(pt)[mcL] >=10^5, BMB <5%. CRi: neutrophils (mcL) <1000 or pt (mcL) <100000, BMB <5%. MLFS: neutrophils (mcL) 1000 and pt (mcL) <10^5, BMB <5%. PR: neutrophils (mcL) >=1000, pt (mcL) >=100000, decrease to 5-25 and >=50% decrease from start. PRi: neutrophils (mcL) <1000 or pt (mcL) <10^5, BMB decrease to 5-25 and >=50% decrease from start. Minor Response: BMB >=25% decrease from start. CRc: neutrophils (mcL) >1,000, pt (mcL) >10^6, BMB <5%. CRm: neutrophils (mcL) >1,000, pt (mcL) >100,000, BMB <5%. For participants with myelodysplastic syndrome (MDS), DMR- CR: >=11 Hgb (g/dL), >=1*10^9 neutrophils(L), >=100*10^9 pt(L), 0% blasts, <=5% BMB. mCR: HI response, <=5% and decreased by >=50% BMB. PR: decrease by >=50% but still >5% BMB. Only those responses which had at least 1 participant were reported.
Time Frame: Day 1 up to end of treatment (maximum up to 486 days)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Participants
  Morphologic CR: AML: number analyzed (Participants) | 4
  Morphologic CR: AML | 1
  Stable disease: AML: number analyzed (Participants) | 4
  Stable disease: AML | 1
  Treatment failure: AML: number analyzed (Participants) | 4
  Treatment failure: AML | 2
  Stable disease: MDS: number analyzed (Participants) | 2
  Stable disease: MDS | 2

56. Secondary Outcome: Number of Participants With Best Response: Combination Cohort 2
Description: Best response observed for: CR, Cri, MLFS, PR, PRi, CRc, CRm. Response criteria for AML- CR:neutrophils(nt)[mcL] >=1000, platelets (mcL) >=100000, BMB <5%. CRi: nt(mcL) <1000 or platelets (mcL) <100000, BMB <5%. MLFS: nt(mcL) 1000 and platelets (mcL) <100000, BMB <5%. PR: nt(mcL) >=1000, platelets (mcL) >=100000, decrease to 5-25 and >=50% decrease from start. PRi: nt(mcL) <1000 or platelets (mcL) <100000, BMB decrease to 5-25 and >=50% decrease from start. Minor Response: BMB >=25% decrease from start. Cytogenetic CR (CRc): nt(mcL) >1,000, platelets (mcL) >100,000, BMB <5%. CRm: nt(mcL) >1,000, platelets (mcL) >100,000, BMB <5%. For participants with myelodysplastic syndrome (MDS), DMR was defined as - CR: >=11 Hgb (g/dL), >=1*10^9 nt(L), >=100*10^9 platelets (L), 0% blasts, <=5% BMB. mCR: HI response, <=5% and decreased by >=50% BMB. PR: decrease by >=50% but still >5% BMB. Only those responses which had at least 1 participant were reported.
Time Frame: Day 1 up to end of treatment (maximum up to 343 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin
Number analyzed (Participants) | 6
Participants
  Morphologic CR: AML | 3
  Morphologic CRi: AML | 2
  MLFs: AML | 2
  PR: AML | 1
  MR: AML | 2
  Treatment failure: AML | 1
  Relapse: AML | 1
  Indeterminate: AML | 1

57. Secondary Outcome: Percentage of Participants With Complete Remission (CR) or CR With Incomplete Blood Count Recovery (CRi) and DMR: Combination Cohort 1
Description: CR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, bone marrow blasts (BMB) <5%. CRi: neutrophils (mcL) <1000 or platelets (mcL) <100000, BMB <5%. DMR included CR, CRi, MLFS, mCR and PR. CR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, bone marrow blasts (BMB) <5%. CRi: neutrophils (mcL) <1000 or platelets (mcL) <100000, BMB <5%. MLFS: neutrophils (mcL) 1000 and platelets (mcL) <100000, BMB <5%. PR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, BMB decrease to 5-25 and >=50% decrease from start.
Time Frame: Day 1 up to end of treatment (maximum up to 486 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Percentage of participants
  CR/CRi | 16.7 [0.4 to 64.1]
  DMR | 16.7 [0.4 to 64.1]

58. Secondary Outcome: Duration of Complete Remission (CR) or CR With Incomplete Blood Count Recovery (CRi) and DMR Response: Combination Cohort 1
Description: Duration of response was the time from the date of first documentation of a CR/CRi and DMR to the date of first documentation of relapse after CR/CRi and DMR or death due to any cause. Duration of response data was censored on the date of the last adequate response assessment for participants who do not have an event (relapse or death). DMR included CR, CRi, MLFS, mCR and PR. CR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, bone marrow blasts (BMB) <5%. CRi: neutrophils (mcL) <1000 or platelets (mcL) <100000, BMB <5%. MLFS: neutrophils (mcL) 1000 and platelets (mcL) <100000, BMB <5%. PR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, BMB decrease to 5-25 and >=50% decrease from start.
Time Frame: Day 1 up to end of treatment (maximum up to 486 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 1
Months
  Duration of CR/CRi | 13.9
  Duration of DMR | 15.3

59. Secondary Outcome: Time to Response: Combination Cohort 1
Description: The time from the date of first dose of study drug to the date of first documentation of a CR or CRi and DMR. DMR included CR, CRi, MLFS, mCR and PR. CR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, BMB <5%. CRi: neutrophils (mcL) <1000 or platelets (mcL) <100000, BMB <5%. MLFS: neutrophils (mcL) 1000 and platelets (mcL) <100000, BMB <5%. PR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, BMB decrease to 5-25 and >=50% decrease from start.
Time Frame: Day 1 up to end of treatment (maximum up to 486 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1. Here, " Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 1
Months
  Time to CR/CRi | 2.1
  Time to DMR | 0.8

60. Secondary Outcome: Overall Survival: Combination Cohort 1
Description: Overall survival was defined as the time from the date of first dose of study drug to the date of death due to any cause. Participants last known to be alive were censored at the date of last contact.
Time Frame: First dose of study drug up to death or date of last contact (maximum up to 514 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg
Number analyzed (Participants) | 6
Months | 11.8 [1.9 to NA] — Upper limit of CI could not be achieved due to less number of participants with event..

61. Secondary Outcome: Overall Survival (OS): Expansion Cohort
Description: OS was defined as the time from the date of first dose of study drug to the date of death due to any cause. Participants last known to be alive were censored at the date of last contact.
Time Frame: First dose of study drug up to death or date of last contact (maximum up to 1408 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 15
Months | 13.6 [3.8 to 18.8]

62. Secondary Outcome: Number of Participants With Best Response: Expansion Cohort
Description: as for outcome 31
Time Frame: From first dose of study drug up to disease progression (maximum duration of 1408 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 15
Participants
  Morphologic CR: AML | 6
  Morphologic CRi: AML | 1
  MLFs: AML | 0
  PR: AML | 0
  PRi: AML | 1
  MR: AML | 2
  SD: AML | 2
  Treatment failure: AML | 2
  Relapse: AML | 0
  Indeterminate: AML | 0
  Not evaluable: AML | 1

63. Secondary Outcome: Percentage of Participants With CR/CRi and DMR: Expansion Cohort
Description: as for outcome 57
Time Frame: Day 1 up to end of treatment (maximum up to 1408 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 15
Percentage of Participants
  Percentage of participants with CR/CRi | 46.7 [21.3 to 73.4]
  Percentage of participants with DMR | 46.7 [21.3 to 73.4]

64. Secondary Outcome: Duration of Response: Expansion Cohort
Description: as for outcome 58
Time Frame: Day 1 up to end of treatment (maximum up to 1408 days)
Population: as for outcome 58
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 7
Months
  Duration of CR/CRi | 9.5 [3.9 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events.
  Duration of DMR | 10.1 [3.9 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

65. Secondary Outcome: Time to Response: Expansion Cohort
Description: as for outcome 59
Time Frame: Day 1 up to end of treatment (maximum up to 1408 days)
Population: as for outcome 58
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 7
Months
  Time to CR/CRi | 5.0 [0.9 to 5.9]
  Time to DMR | 2.3 [0.9 to 5.0]

66. Secondary Outcome: Ratio of GLI1 Levels at Baseline to Day 21 Cycle 1: Expansion Cohort
Description: Biomarker assessments were used to understand the in vivo mechanism of action of PF-04449913, as well as potential mechanisms of resistance. In this outcome measure ratio of GLI1 levels (Blood, mRNA) at baseline to day 21 cycle 1 is reported.
Time Frame: Baseline, Day 21 of Cycle 1(Predose)
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 3
Ratio | 0.905 (0.4147)

67. Secondary Outcome: Multiple Dose- Cmax, Cmin, Cavg, and Ctrough of PF-04449913: Combination Cohort 3
Description: as for outcome 24
Time Frame: Cmax, Cmin: Pre-dose, 0.25, 1, 4, 6, 24 hours post PF-04449913 dosing on Day 7 and Day 21 of Cycle 1; Cavg: 0 to 24 hors post PF-04449913 dosing on Day 7 and Day 21 of Cycle 1; Ctrough: Pre PF-04449913 dosing on Day 7 and Day 21 of Cycle 1
Population: as for outcome 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Nanogram per milliliter
  Cmax: Cycle 1/Day 7: number analyzed (Participants) | 5
  Cmax: Cycle 1/Day 7 | 1387 (22)
  Cmin: Cycle 1/Day 7: number analyzed (Participants) | 5
  Cmin: Cycle 1/Day 7 | 414.1 (33)
  Cavg: Cycle 1/Day 7: number analyzed (Participants) | 5
  Cavg: Cycle 1/Day 7 | 834.6 (22)
  Ctrough: Cycle 1/Day 7: number analyzed (Participants) | 5
  Ctrough: Cycle 1/Day 7 | 526.3 (28)
  Cmax: Cycle 1/Day 21 | 1218 (51)
  Cmin: Cycle 1/Day 21 | 323.2 (46)
  Cavg: Cycle 1/Day 21 | 701.9 (44)
  Ctrough: Cycle 1/Day 21 | 347.5 (45)

68. Secondary Outcome: Multiple Dose- Tmax of PF-04449913: Combination Cohort 3
Time Frame: Pre-dose, 0.25, 1, 4, 6, 24 hours post PF-04449913 dosing on Day 7 and Day 21 of Cycle 1
Population: as for outcome 36
Measure: Median (Full Range); unit: Hours
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Hours
  Cycle 1/Day 7: number analyzed (Participants) | 5
  Cycle 1/Day 7 | 4.000 [3.90 to 6.00]
  Cycle 1/Day 21 | 2.500 [0.900 to 5.98]

69. Secondary Outcome: Multiple Dose- AUCtau of PF-04449913: Combination Cohort 3
Description: AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours.
Time Frame: 0 to 24 hours post PF-04449913 dosing on Day 7 and Day 21 of Cycle 1
Population: as for outcome 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Nanogram*hour per milliliter
  Cycle 1/Day 7: number analyzed (Participants) | 5
  Cycle 1/Day 7 | 20010 (22)
  Cycle 1/Day 21 | 16860 (44)

70. Secondary Outcome: Multiple Dose- CL/F of PF-04449913: Combination Cohort 3
Description: as for outcome 22
Time Frame: Pre-dose, 0.25, 1, 4, 6, 24 hours post PF-04449913 dosing on Day 7 and Day 21 of Cycle 1
Population: as for outcome 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Liter per hour
  Cycle 1/Day 7: number analyzed (Participants) | 5
  Cycle 1/Day 7 | 4.999 (22)
  Cycle 1/Day 21 | 5.936 (44)

71. Secondary Outcome: Multiple Dose- Cmax, Cmin, Cavg, and Ctrough of Azacitidine: Combination Cohort 3
Description: Cmax = Maximum plasma concentration, observed directly from data. Cmin = Minimum plasma concentration observed directly from data. Cavg = Average plasma concentration over the dosing interval of 24 hours. Ctrough = Pre-dose concentration, observed directly from data.
Time Frame: Cmax: 0.25, 0.5, 1, 2, 6 hrs post azacitidine dose on Day 1/Cycle 1;Cmin: Pre-dose, 0.25, 0.5, 1, 2, 6 hrs post azacitidine dose on Day 7/Cycle 1;Cavg: 0 to 24 hrs post azacitidine dose on Day 7/Cycle 1;Ctrough:Pre azacitidine dose on Day 7/Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Nanogram per milliliter
  Cmax: Cycle 1/Day 1 | 1803 (60)
  Cmax: Cycle 1/Day 7 | 1717 (49)
  Cmin: Cycle 1/Day 7 | NA (NA) — Cmin was not estimable as the analyte was not detected for any participant.
  Cavg: Cycle 1/Day 7 | 51.60 (30)
  Ctrough: Cycle 1/Day 7 | NA (NA) — Ctrough was not estimable as the analyte was not detected for any participant.

72. Secondary Outcome: Multiple Dose- Tmax of Azacitidine: Combination Cohort 3
Time Frame: 0.25, 0.5, 1, 2, and 6 hours post azacitidine dosing on Day 1 of Cycle 1 and pre-dose, 0.25, 0.5, 1, 2, and 6 hours post azacitidine dosing on Day 7 of Cycle 1
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Hours
  Day 1 | 0.2500 [0.233 to 0.500]
  Day 7 | 0.2500 [0.233 to 0.500]

73. Secondary Outcome: Multiple Dose- AUCtau and AUCinf of Azacitidine: Combination Cohort 3
Description: AUCtau, was determined by linear/log trapezoidal method. For AUC, tau (dosing interval) was 24 hours. AUCinf = AUClast + (Clast/kel), where Clast = predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and where kel = terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: AUCinf: 0.25, 0.5, 1, 2, and 6 hours post azacitidine dosing at Day 1 of Cycle 1 and pre-dose, 0.25, 0.5, 1, 2, and 6 hours post azacitidine dosing at 7 of Cycle 1; AUCtau: 0 to 24 hours post azacitidine dosing on Day 1 and 7 of Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Nanogram*hour per milliliter
  AUCtau: Cycle 1/Day 1 | 1200 (28)
  AUCinf: Cycle 1/Day 1 | 910.9 (39)
  AUCtau: Cycle 1/Day 7 | 1241 (30)
  AUCinf: Cycle 1/Day 7 | 1200 (33)

74. Secondary Outcome: Overall Survival: Combination Cohort 3
Description: as for outcome 60
Time Frame: First dose of study drug up to death or date of last contact (maximum up to 841 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Months | 30.3 [6.1 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

75. Secondary Outcome: Ratio of GLI1 Levels at Baseline to End of Treatment: Combination Cohort 3
Description: Biomarker assessments were used to understand the in vivo mechanism of action of PF-04449913, as well as potential mechanisms of resistance. In this outcome measure ratio of GLI1 levels (Blood, mRNA) to end of treatment is reported.
Time Frame: Baseline, at the end of treatment (hours unspecified, any day maximum up to 841 days)
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 1
Ratio | 0.776 (NA) — Standard deviation could not be estimated as there was only 1 participant evaluable.

76. Secondary Outcome: Number of Participants With Best Response: Combination Cohort 3
Description: Best response observed for: CR, Cri, MLFS, PR, PRi, CRc, CRm. Response criteria for participants with AML- CR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, BMB <5%. CRi: neutrophils (mcL) <1000 or platelets (mcL) <100000, BMB <5%. MLFS: neutrophils (mcL) 1000 and platelets (mcL) <100000, BMB <5%. PR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, decrease to 5-25 and >=50% decrease from start. PRi: neutrophils (mcL) <1000 or platelets (mcL) <100000, BMB decrease to 5-25 and >=50% decrease from start. Minor Response: BMB >=25% decrease from start. CRc: neutrophils (mcL) >1,000, platelets (mcL) >100,000, BMB <5%. CRm: neutrophils (mcL) >1,000, platelets (mcL) >100,000, BMB <5%. Only those responses which had at least 1 participant were reported.
Time Frame: Day 1 up to end of treatment (maximum up to 841 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Participants
  Morphologic CR | 3
  PRi | 1
  Treatment failure | 2

77. Secondary Outcome: Percentage of Participants With CR/CRi and DMR: Combination Cohort 3
Description: as for outcome 57
Time Frame: Day 1 up to end of treatment (maximum up to 841 days)
Population: FAS included all enrolled participants who received at least 1 dose of study medication on or after Cycle 1/Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 6
Percentage of participants
  CR/Cri: number analyzed (Participants) | 3
  CR/Cri | 50.0 [11.8 to 88.2]
  DMR: number analyzed (Participants) | 3
  DMR | 50.0 [11.8 to 88.2]

78. Secondary Outcome: Duration of Complete Remission (CR) or CR With Incomplete Blood Count Recovery (CRi) and DMR Response: Combination Cohort 3
Description: as for outcome 58
Time Frame: Day 1 up to end of treatment (maximum up to 841 days)
Population: as for outcome 58
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 3
Months
  Duration of CR/CRi | 6.6 [5.6 to 11.1]
  Duration of DMR | 6.6 [5.6 to 19.8]

79. Secondary Outcome: Time to Complete Remission (CR) or CR With Incomplete Blood Count Recovery (CRi) and DMR Response: Combination Cohort 3
Description: The time from the date of first dose of study drug to the date of first documentation of a CR or CRi and DMR. DMR included CR, CRi, MLFS, mCR and PR. CR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, bone marrow blasts (BMB) <5%. CRi: neutrophils (mcL) <1000 or platelets (mcL) <100000, BMB <5%. MLFS: neutrophils (mcL) 1000 and platelets (mcL) <100000, BMB <5%. PR: neutrophils (mcL) >=1000, platelets (mcL) >=100000, BMB decrease to 5-25 and >=50% decrease from start.
Time Frame: Day 1 up to end of treatment (maximum up to 841 days)
Population: as for outcome 58
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Cohort 3: PF-04449913 100 mg + Azacitidine
Number analyzed (Participants) | 3
Months
  Time to CR/CRi | 5.9 [5.8 to 11.5]
  Time to DMR | 5.8 [2.8 to 5.9]

80. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities: Continuation Cohort
Description: Laboratory parameters included- hematology: lymphocytes/leukocytes (%), neutrophils/leukocytes (%), basophils/leukocytes (%), eosinophils/leukocytes (%), monocytes/leukocytes (%), prothrombin time (sec), blasts/leukocytes (%); clinical chemistry: lactate dehydrogenase (u/l), protein (g/l), blood urea nitrogen (BUN) (mmol/l), urate (mmol/l), chloride (mmol/l), calcium (mmol/l); urinalysis: specific gravity (scalar), pH (scalar), urine glucose (scalar), ketones (scalar), nitrite, leukocyte esterase, urine erythrocytes (scalar), urine leukocytes (scalar). In this outcome measure participants for each laboratory parameter were evaluated as normal, abnormal low only, abnormal high only or abnormal low and an abnormal high. Laboratory values were as per laboratory normal ranges. Values above normal range = abnormal high and below range = abnormal low. Participants with both an abnormal low and an abnormal high value while on study were reported as 'Abnormal low and Abnormal high'.
Time Frame: Baseline up to maximum 1146 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication. Here, "Number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg
Number analyzed (Participants) | 1
Participants | 0

81. Secondary Outcome: Number of Participants With TEAEs, Serious TEAEs, Treatment Related TEAEs, Grade 3 or 4 TEAEs Based on NCI CTCAE v4.0: Expansion Cohort
Description: AE:any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Serious AE:any untoward medical occurrence at any dose that resulted in death,was life threatening,required inpatient hospitalization or prolongation of existing hospitalization;resulted in persistent or significant disability/incapacity,resulted in congenital anomaly/birth defect. TEAEs:events absent before treatment or that worsened relative to pretreatment state. Treatment-related TEAE:any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to drug was assessed by the Investigator. National cancer institute common terminology criteria (NCI-CTCAE) Grade(G) v4.0:G 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; G 4:life-threatening consequence, urgent intervention indicated.
Time Frame: Day 1 up to 28 days after last dose of study drug (Maximum up to 1436 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 15
Participants
  TEAEs | 15
  Serious TEAEs | 9
  Treatment related TEAEs | 14
  Grade 3 or 4 TEAEs | 12

82. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs: Expansion Cohort
Description: Vital signs included blood pressure (sitting or supine) and heart rate. Vital sign criteria included: Systolic BP: <90 millimeter of mercury [mmHg]; Systolic BP change from baseline: maximum increase and decrease >=30 mmHg; Diastolic BP minimum < 50 mmHg; Diastolic BP change from baseline: maximum decrease and increase >=20 mmHg; heart rate <40 and >120 beats per minute. Clinically significant changes in vital signs were determined by the investigator's discretion.
Time Frame: Baseline up to maximum 1436 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 15
Participants | 0

83. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs: Continuation Cohort
Description: as for outcome 82
Time Frame: Baseline up to maximum 1146 days
Population: as for outcome 80
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg
Number analyzed (Participants) | 1
Participants | 0

84. Secondary Outcome: Number of Participants With TEAEs, Serious TEAEs, Treatment Related TEAEs, Grade 3 or 4 TEAEs Based on NCI CTCAE v4.0: Continuation Cohort
Description: AE: any untoward medical occurrence in participant who received study drug or medical device without regard to possibility of causal relationship with the treatment or usage. Serious AE: any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. TEAEs: events absent before treatment or that worsened relative to pretreatment state. Treatment-related TEAE: any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to drug was assessed by the Investigator. NCI-CTCAE Grade: Grade 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4= life-threatening consequence, urgent intervention indicated.
Time Frame: Day 1 up to 28 days after last dose of study drug (Maximum up to 1146 days)
Population: as for outcome 80
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg
Number analyzed (Participants) | 1
Participants
  TEAEs | 1
  Serious TEAEs | 0
  Treatment Related TEAEs | 1
  Grade 3 or 4 TEAEs | 0

85. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities: Expansion Cohort
Description: as for outcome 80
Time Frame: Baseline up to maximum 1436 months
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after last dose of study drug. Monotherapy cohort, a) 25 mg: maximum up to 136 days; b) 50 mg: maximum up to 179 days; c) 100 mg: maximum up to 472 days. Combination cohort 1: maximum up to 514 days. Combination cohort 2: maximum up to 371 days. Combination cohort 3: maximum up to 869 days. Expansion cohort: maximum up to 1436 days. Continuation cohort: Maximum up to 1146 days.
Arm/Group | Monotherapy Cohort: PF-04449913 (Glasdegib) 25 mg | Monotherapy Cohort: PF-04449913 50 mg | Monotherapy Cohort: PF-04449913 100 mg | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin | Combination Cohort 3: PF-04449913 100 mg + Azacitidine | Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/4 | 0/6 | 5/6 | 2/6 | 4/6 | 0/1 | 11/15
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/4 | 1/6 | 1/6 | 4/6 | 1/6 | 0/1 | 9/15
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 6/6 | 6/6 | 6/6 | 1/1 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy Cohort: PF-04449913 (Glasdegib) 25 mg (N=3) | Monotherapy Cohort: PF-04449913 50 mg (N=4) | Monotherapy Cohort: PF-04449913 100 mg (N=6) | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg (N=6) | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin (N=6) | Combination Cohort 3: PF-04449913 100 mg + Azacitidine (N=6) | Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg (N=1) | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy Cohort: PF-04449913 (Glasdegib) 25 mg (N=3) | Monotherapy Cohort: PF-04449913 50 mg (N=4) | Monotherapy Cohort: PF-04449913 100 mg (N=6) | Combination Cohort 1 (Unfit Participants): PF-04449913 100 mg + LDAC 20 mg (N=6) | Combination Cohort 2 (Fit Participants): PF-04449913 100 mg + Cytarabine + Daunorubicin (N=6) | Combination Cohort 3: PF-04449913 100 mg + Azacitidine (N=6) | Continuation Cohort (Monotherapy Cohort): PF-04449913 100 mg (N=1) | Expansion Cohort (Unfit Participants): PF-04449913 100 mg+ LDAC 20 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3 | 4 | 2 | 0 | 10
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 4 | 2 | 0 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 6 | 3 | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 5 | 2 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 2 | 6 | 3 | 0 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 3 | 2 | 2 | 1 | 1 | 6
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 4 | 5 | 0 | 10
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 4
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Malaise (General disorders) | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 2
Medical device site ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 2 | 2 | 3 | 2 | 1 | 7
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 7
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 3
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 2
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood zinc decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4
Platelet count decreased (Investigations) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 7
Weight decreased (Investigations) | 0 | 2 | 1 | 2 | 3 | 2 | 0 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 3 | 1 | 4 | 2 | 0 | 7
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 3 | 0 | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Cytarabine syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 0 | 1 | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 3 | 5 | 4 | 5 | 3 | 0 | 6
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 3 | 1 | 0 | 3
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Auricular chondritis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infective tenosynovitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibrin degradation products increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT02038777/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT02038777/SAP_001.pdf